CLINICAL TRIAL: NCT06939660
Title: Spatiotemporal Spinal Cord Stimulation Based on Implantable Brain-machine Interfaces and Exoskeletons for Spinal Cord Injury (BASEGO)
Brief Title: BCI-Assisted SCS-EXS for Gait Optimization
Acronym: BASEGO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Beijing Xinzhida Neural Technology Co., Ltd (Unknown); Beijing Pins Medical Co., Ltd (Industry); Hangzhou RoboCT Technology Development Co.,Ltd (Unknown)
Responsible Party: Principal Investigator, Wanru Duan, Chief physician, Xuanwu Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRWEP2024W022010200-SCS01
Record Dates: First submitted 2025-04-02; First posted 2025-04-23 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Spinal Cord Injuries (SCI); Spinal Cord Injury, Chronic; Spinal Cord Injury; Spinal Cord Injury Cervical; Spinal Cord Injury Thoracic; Spinal Cord Injury (Quadraplegia); Motor Impairment; Motor Deficits; Gait Training; Gait Impairment
Keywords: Brain-computer interface; Spianl cord stimulation; Exoskeleton; Rehabilitation; Spinal cord injury; Motor dysfunction; BCI; Brain-spinal interface; BSI; Brain-machine interface; Gait training; Neural plasticity
MeSH Terms: conditions — Spinal Cord Injuries; Bronchiolitis Obliterans Syndrome; Quadriplegia; Neurologic Manifestations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCI-SCS-EXO (Experimental): Participants will undergo a BCI-SCS-EXS intervention, involving implatation of high-density ECoG electrodes, as well as SCS electrodes. The system will be calibrated to synchronize BCI-decoded motor intent with SCS parameters and integrate with the exoskeleton (EXS) to provide synchronized gait assistance. Safety and efficacy assessments will be conducted at 1, 2, 3, 6, and 12 months post-intervention.
  Interventions: Device: BCI-SCS-EXS

INTERVENTIONS:
Device: BCI-SCS-EXS — Participants will undergo a BCI-SCS-EXS intervention designed to enhance neurorehabilitation for spinal cord injury (SCI). The intervention includes:
  1. BCI Implantation: High-density ECoG electrodes placed over the motor cortex to decode lower limb movement intent.
  2. SCS Electrode Implantation: 5-6-5 paddle electrodes implanted at T11-L2 to deliver targeted spinal cord stimulation.
  3. System Calibration: BCI-SCS synchronization to trigger stimulation parameters based on decoded motor intent. SCS-EXS integration to provide synchronized gait assistance.
  4. Rehabilitation Training: Daily training sessions (60 minutes, 5 times/week for 1 year) combining BCI-SCS-EXS.
  5. Follow-Up: Safety and efficacy assessments at 1, 2, 3, 6, and 12 months post-intervention.
  This intervention aims to promote neuroplasticity and functional recovery through brain-controlled spinal activation and synchronized exoskeleton assistance.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and technical feasibility of a novel brain-machine interface (BCI)-assisted spinal cord stimulation (SCS) and exoskeleton (EXS) system in patients with spinal cord injury (SCI). The primary aim is to determine whether the BCI-SCS-EXS system can safely and effectively improve lower limb motor function and quality of life in individuals with chronic SCI.

Participant Population:

Adults aged 14-65 years (sex/gender not limited). Patients with chronic SCI (≥6 months post-injury) classified as ASIA A, B, or C.

Individuals with stable health status, MMSE ≥22, and secondary education or above.

Primary Questions:

1. Is the BCI-SCS-EXS system safe and technically feasible for SCI rehabilitation?
2. Does the system improve lower limb motor function and quality of life in SCI patients?

Interventions:

Participants will undergo the following procedures:

Phase I (Implantation):

BCI implantation: ECoG electrodes placed over the motor cortex to decode lower limb movement intent.

SCS electrode implantation: 5-6-5 paddle electrodes at T11-L2 for targeted spinal cord stimulation.

Phase II (System Calibration):

BCI-SCS synchronization: Calibration of decoded motor intent to trigger SCS parameters.

SCS-EXO synchronization: Integration of SCS pulses with exoskeleton-assisted gait training.

Phase III (Rehabilitation):

Daily BCI-SCS-EXS training sessions (60 minutes, 5 times/week for 1 year). Adaptive adjustments to stimulation parameters and exoskeleton support based on performance.

Remote monitoring of device performance and emergency intervention for technical issues.

Outcome Measures:

Primary: Safety (adverse events, device performance, synchronization metrics). Secondary: Efficacy (motor function, neurophysiological function, quality of life).

Ethics and Safety:

Informed consent will be obtained from all participants. Adverse events will be monitored and reported according to CTCAE 5.0 guidelines.

Participant confidentiality will be strictly maintained. This study will provide foundational evidence for the safety and feasibility of the BCI-SCS-EXO system, paving the way for future randomized controlled trials in SCI rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Age 14-65 years, any gender.
* Clinical diagnosis of spinal cord injury (SCI) due to trauma, inflammation, tumor, vascular disease, or iatrogenic factors, confirmed by medical history, physical examination, and ancillary tests, resulting in lower limb motor dysfunction.
* SCI diagnosed ≥6 months prior, with ≥1 month of continuous conventional rehabilitation (e.g., physical therapy, acupuncture, hydrotherapy, ≥3 hours daily) without significant improvement in motor function in the past 2 months.
* ASIA Impairment Scale (AIS) grade A, B, or C based on the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI).
* Good general health with a life expectancy ≥12 months.
* Mini-Mental State Examination (MMSE) score ≥22.
* Educational attainment of secondary school or above.
* Willingness to participate, provide informed consent, and comply with study follow-up.

Exclusion Criteria:

* Presence of diseases other than spinal cord injury (SCI) that affect lower limb motor function, including brain diseases (e.g., brain tumor, stroke), lower limb vascular diseases (e.g., lower limb vascular occlusion), peripheral nerve diseases, or lower limb bone diseases (e.g., osteoarthritis, joint contracture).
* Requires continuous medical interventions (e.g., tracheal intubation, nasogastric feeding) to maintain critical physiological functions (e.g., heartbeat, respiration, swallowing).
* Congenital or acquired structural abnormalities of the lower limb bones or muscles.
* Presence of surgical contraindications (e.g., anesthesia-related adverse reactions, coagulation risks, or surgeon's determination of unsuitability for surgery).
* Presence of active implantable devices except for SCS or BCI devices (e.g., pacemakers, defibrillators, drug infusion pumps, cochlear implants, sacral nerve stimulators).
* Unable to receive implantable devices due to other disease treatments or investigations, or requires magnetic resonance imaging (MRI) during the device implantation period.
* MRI shows structural damage >50% in motor function areas (precentral and postcentral gyri, ventromedial sensorimotor areas, mid temporal lobe, Broca's area, Wernicke's area, Geschwind's area), or DTI shows damage >50% in the posterior limb of the internal capsule.
* Severe cardiovascular disease: Above level II myocardial ischemia or myocardial infarction, uncontrolled arrhythmias (including QTc interval ≥450 ms in men, ≥470 ms in women), level III-IV heart failure (NYHA classification), or echocardiography showing LVEF <50%.
* Coagulation abnormalities (INR >1.5 ULN, PT >ULN +4 s, or APTT >1.5 ULN), hemorrhagic tendency, or undergoing thrombolytic or anticoagulant therapy.
* Severe infections within 4 weeks before surgery (requiring IV antibiotics, antifungals, or antivirals) or lumbar soft tissue infections, or unexplained fever >38.5℃ during screening or before surgery.
* HIV infection, acquired immunodeficiency syndrome (AIDS), active tuberculosis, active hepatitis B (HBV DNA ≥500 IU/ml), hepatitis C (positive HCV antibody and detectable HCV-RNA), or co-infection of hepatitis B and C.

Severe cerebrovascular events (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, or pulmonary embolism within 12 months before enrollment.

* Metastatic malignancies or untreated malignant tumors.
* Major surgery or severe traumatic injuries, fractures, or ulcers within 4 weeks before enrollment.
* Addictive habits such as drug abuse or alcoholism.
* History of psychotropic drug abuse that is not controllable or presence of mental disorders, including major psychiatric illnesses (e.g., depression [BDI score >20], anxiety, obsessive-compulsive disorder, schizophrenia, autism, chronic sleep disorders, consciousness disorders).
* Pregnant, breastfeeding, planning to conceive, or women of childbearing potential without reliable contraception.
* Participation in other clinical trials within the past month.
* Cognitive impairments or poor compliance from subjects, family members, or caregivers, or inability to complete at least 12 months of follow-up and rehabilitation training.
* Other conditions that increase the risk of study participation or device use, as determined by the investigator.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
The content and number of AEs as well as their severity according to CTCAE v6.0 | 0-12 months post-implantation
  The safety of the BCI-SCS-EXS system is evaluated by focusing on adverse events (AEs) associated with the trial devices (BCI, SCS, and EXS). AEs are documented and categorized according to their severity and relationship to the devices. The primary outcome measure calculated as the content and number of AEs as well as their severity according to CTCAE v6.0. This metric provides an overview of the safety profile of the BCI-SCS-EXS system.

SECONDARY OUTCOMES:
Signal Acquisition Normal Rate of BCI | 0, 1, 2, 3, 6, 12 months post-implantation
  Signal Acquisition Normal Rate is quantified as the ratio of successfully captured high-quality ECoG signal segments to the total number of predefined-length segments. This metric is calculated by analyzing the proportion of segments that meet predefined quality criteria as signal-to-noise ratio (SNR) >10 dB. The rate is expressed as a percentage and reflects the reliability of the BCI system in capturing usable signals.
Electrode Impedance of BCI electrodes | 0, 1, 2, 3, 6, 12 months post-implantation
  Electrode impedance is measured to ensure optimal signal transmission. Impedance is assessed using an EEG acquisition system with a low-noise preamplifier and impedance detection software. The impedance value, expressed in kilohms (kΩ), reflects the resistance between the electrode and scalp.
Effective Channel Count of BCI | 0, 1, 2, 3, 6, 12 months post-implantation
  The effective channel count is quantified by the number of channels with a signal-to-noise ratio (SNR) exceeding 10 dB. SNR is calculated by analyzing the power spectral density of each channel. The count reflects the system's ability to reliably capture high-quality neural signals.
Electrode Impedance Stability of SCS | 0, 1, 2, 3, 6, 12 months post-implantation
  Electrode impedance stability is assessed by measuring the impedance of each SCS electrode channel at regular intervals. Impedance is measured using a calibrated impedance meter integrated with the SCS system. The stability is quantified by calculating the coefficient of variation (CV) of impedance values over time. A lower CV indicates more stable impedance.
Position Stability of SCS | 0, 3, 6, 12 months post-implantation
  Position stability is evaluated using X-ray imaging to confirm the placement of SCS electrodes relative to the T12 vertebral body. Stability is quantified by comparing the initial position with subsequent measurements over time. A positional shift greater than 2 mm is considered significant, indicating potential instability.
Battery Fault Rate of SCS | 0-12 months post-implantation
  The battery fault rate is quantified by recording the number of unexpected battery failures or shutdowns during the study period. This metric is calculated as the total count of such events divided by the total number of battery operation days. The rate is expressed as a percentage to reflect the reliability of the SCS system's power supply over time.
Command Trigger Success Rate of BCI-SCS Matching | 0, 1, 2, 3, 6, 12 months post-implantation
  The command trigger success rate is quantified as the percentage of BCI commands that successfully activate the SCS system. This is calculated as dividing the number of successful triggers by the total number of BCI commands issued during 5 minutes. The rate is expressed as a percentage, with higher values indicating more reliable BCI-SCS synchronization.
Delay Drift Deviation of BCI-SCS Matching | 0, 1, 2, 3, 6, 12 months post-implantation
  The delay drift deviation is quantified by measuring the temporal deviation of the actual delay between BCI command issuance and SCS response from the intended delay. This deviation is calculated as the average difference in milliseconds over a 5-minute trial. Lower values indicate more precise synchronization between the BCI and SCS systems.
Recognition Accuracy of BCI Brain Signal Decoding | 0, 1, 2, 3, 6, 12 months post-implantation
  The recognition accuracy is quantified through offline analysis using confusion matrices to evaluate the precision of movement intent decoding. Accuracy is calculated as the ratio of correctly decoded commands to the total number of commands analyzed, expressed as a percentage. Higher accuracy values indicate more reliable BCI signal decoding.
Latency of BCI Brain Signal Decoding | 0, 1, 2, 3, 6, 12 months post-implantation
  The latency is quantified as the time interval from the acquisition of ECoG signals to the generation of control commands. This is measured in milliseconds using timestamp synchronization between signal capture and command output. Lower latency values indicate more efficient real-time decoding performance of the BCI system.
Gait Trigger Delay of SCS-EXS Matching | 0, 1, 2, 3, 6, 12 months post-implantation
  The gait trigger delay is quantified as the time interval from the initiation of an SCS pulse to the commencement of exoskeleton joint movement. This delay is measured using synchronized data logging from both the SCS device and the exoskeleton's motion sensors, with the time difference calculated in milliseconds. Lower values indicate more precise synchronization between spinal cord stimulation and exoskeleton-assisted gait.
Joint Movement Consistency of SCS-EXS Matching | 0, 1, 2, 3, 6, 12 months post-implantation
  The joint movement consistency is quantified by measuring the correlation between hip/knee/ankle joint movements and SCS stimulation pulses using Pearson correlation coefficients. Joint movements are captured via motion sensors, while SCS pulses are logged by the stimulation device. The Pearson coefficient is calculated for each joint, with values closer to +1 or -1 indicating stronger consistency between joint movement and stimulation timing.
Lower Limb Motor Score (LEMS) | 0, 1, 2, 3, 6, 12 months post-implantation
  The LEMS quantifies motor function recovery of key muscle groups in the lower limbs by assessing muscle strength on a scale from 0 (no movement) to 5 (normal strength) for each muscle group. The total score is calculated by summing the individual muscle scores of iliopsoas, quadriceps femoris, and tibialis anterior muscles, with higher scores indicating better motor function recovery.
Muscle Strength of Lower Limbs | 0, 1, 2, 3, 6, 12 months post-implantation
  Muscle strength is assessed using the Medical Research Council (MRC) grading scale for the iliopsoas, quadriceps femoris, gastrocnemius, and tibialis anterior muscles. The MRC scale ranges from 0 to 5, with 0 indicating no muscle contraction and 5 indicating normal strength. Each muscle group is evaluated individually, and the scores are recorded to quantify the strength of each muscle. Higher MRC grades indicate better muscle function.
Assisted Standing Time | 0, 1, 2, 3, 6, 12 months post-implantation
  Assisted standing time is quantified as the duration patients can stand independently with exoskeleton assistance. This is measured in seconds using a stopwatch or timing software. The assessment is conducted in a standardized environment to ensure consistency. Longer durations indicate improved standing endurance and stability.
10-Meter Walk Test (10MWT) | 0, 1, 2, 3, 6, 12 months post-implantation
  The 10MWT measures walking or assisted walking speed over a 10-meter distance. Walking speed is calculated by timing the duration it takes for a patient to walk 10 meters at their comfortable pace. The speed is then expressed in meters per second (m/s). Higher walking speeds indicate better mobility and functional recovery.
Gait Step Length | 0, 1, 2, 3, 6, 12 months post-implantation
  These metrics are captured using motion analysis systems. Step length is measured in centimeters during 10MWT. Higher step length indicate improved walking function.
Gait Joint Range | 0, 1, 2, 3, 6, 12 months post-implantation
  These metrics are captured using motion analysis systems. Joint range of motion is measured in degrees during 10MWT. Higher joint range of motion indicate improved walking function.
Gait Symmetry | 0, 1, 2, 3, 6, 12 months post-implantation
  These metrics are captured using motion analysis systems. Gait Symmetry is measured during 10MWT by comparing the consistency of steps between limbs. More symmetrical gait patterns, indicate improved walking function.
Surface Electromyography (sEMG) | Time frame: 0, 1, 2, 3, 6, 12 months post-implantation
  sEMG measures resting and task-specific muscle activity during leg and knee extension. Muscle activity is captured using surface electrodes placed over target muscles, with signals recorded in microvolts (µV). Activity is quantified by calculating the root mean square (RMS) of the signal over a defined period. Higher RMS values indicate greater muscle activation during specific tasks.
Nerve Conduction Velocity | 0, 6, 12 months post-implantation
  Nerve conduction velocity is quantified via EMG to assess the efficiency of neural signal transmission in limb muscles. This involves stimulating specific nerves and recording the resulting muscle action potentials. The conduction velocity is calculated by measuring the distance between the stimulation point and the recording electrode, divided by the latency of the evoked response, expressed in meters per second (m/s). Higher values indicate more efficient nerve conduction.
Urodynamics | 0, 6, 12 months post-implantation
  Urodynamics is quantified by measuring bladder residual volume and maximum free urine flow rate. Bladder residual volume is assessed using ultrasound or catheterization, expressed in milliliters (mL). Maximum free urine flow rate is measured during spontaneous voiding, expressed in milliliters per second (mL/s). These parameters provide insights into bladder function and urinary tract efficiency.
SF-36 Health Survey | 0, 1, 2, 3, 6, 12 months post-implantation
  The SF-36 Health Survey quantifies physical and mental health-related quality of life through a standardized questionnaire. This survey includes multiple domains such as physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. Each domain is scored on a scale from 0 to 100, with higher scores indicating better health status and quality of life.
SCI-QOL Psychological Adaptation Subscale | 0, 1, 2, 3, 6, 12 months post-implantation
  The SCI-QOL Psychological Adaptation Subscale quantifies psychological adaptation to spinal cord injury (SCI) through a series of Likert-scale items. This subscale assesses various aspects of psychological well-being, including emotional well-being, depression, anxiety, stigma, grief/loss, self-evaluation, and psychological trauma. Each item is scored on a scale from 1 to 5, with higher scores indicating better psychological adaptation and mental health.
Cognitive Function by MMSE | 0, 1, 2, 3, 6, 12 months post-implantation
  The Mini-Mental State Examination (MMSE) evaluates orientation, registration, attention, recall, and language, with scores ranging from 0 to 30, where higher scores indicate better cognitive function.
Cognitive Function by MoCA | 0, 1, 2, 3, 6, 12 months post-implantation
  The Montreal Cognitive Assessment (MoCA) assesses a broader range of cognitive domains, including attention, executive function, memory, language, visuospatial abilities, and abstraction, with scores ranging from 0 to 30. Higher scores on both tests indicate better cognitive performance.
Pain Intensity | 0, 1, 2, 3, 6, 12 months post-implantation
  Pain intensity is quantified using the Visual Analog Scale (VAS). Patients are asked to rate their pain on a continuous scale from 0 to 10, where 0 represents no pain and 10 represents the worst possible pain. The score is recorded in numerical values, with lower scores indicating less pain intensity.
Psychosocial Impact of Assistive Devices | 0, 1, 2, 3, 6, 12 months post-implantation
  The psychosocial impact of assistive devices is evaluated using the Psychosocial Impact of Assistive Devices Scale (PIADS). This scale assesses the influence of assistive devices on an individual's competence, adaptability, and self-esteem. Each domain is scored on a scale from -3 to +3, with higher positive scores indicating a more favorable impact on psychosocial well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital ,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the inclusion of proprietary and commercially sensitive information related to the development and operation of the BCI-SCS-EXS system. The data contain technical specifications, algorithmic details, and performance metrics that are protected as intellectual property by the collaborating research institutions and industry partners. Sharing such data could compromise competitive advantages, hinder future innovation, and violate confidentiality agreements. However, aggregated and anonymized results will be made available upon reasonable request for scientific and regulatory purposes, ensuring transparency while safeguarding commercial interests.

REFERENCES:
- [Background] Gad P, Gerasimenko Y, Zdunowski S, Turner A, Sayenko D, Lu DC, Edgerton VR. Weight Bearing Over-ground Stepping in an Exoskeleton with Non-invasive Spinal Cord Neuromodulation after Motor Complete Paraplegia. Front Neurosci. 2017 Jun 8;11:333. doi: 10.3389/fnins.2017.00333. eCollection 2017. PMID 28642680
- [Background] Gorgey AS, Gill S, Holman ME, Davis JC, Atri R, Bai O, Goetz L, Lester DL, Trainer R, Lavis TD. The feasibility of using exoskeletal-assisted walking with epidural stimulation: a case report study. Ann Clin Transl Neurol. 2020 Feb;7(2):259-265. doi: 10.1002/acn3.50983. Epub 2020 Feb 5. PMID 32023011
- [Background] Rowald A, Komi S, Demesmaeker R, Baaklini E, Hernandez-Charpak SD, Paoles E, Montanaro H, Cassara A, Becce F, Lloyd B, Newton T, Ravier J, Kinany N, D'Ercole M, Paley A, Hankov N, Varescon C, McCracken L, Vat M, Caban M, Watrin A, Jacquet C, Bole-Feysot L, Harte C, Lorach H, Galvez A, Tschopp M, Herrmann N, Wacker M, Geernaert L, Fodor I, Radevich V, Van Den Keybus K, Eberle G, Pralong E, Roulet M, Ledoux JB, Fornari E, Mandija S, Mattera L, Martuzzi R, Nazarian B, Benkler S, Callegari S, Greiner N, Fuhrer B, Froeling M, Buse N, Denison T, Buschman R, Wende C, Ganty D, Bakker J, Delattre V, Lambert H, Minassian K, van den Berg CAT, Kavounoudias A, Micera S, Van De Ville D, Barraud Q, Kurt E, Kuster N, Neufeld E, Capogrosso M, Asboth L, Wagner FB, Bloch J, Courtine G. Activity-dependent spinal cord neuromodulation rapidly restores trunk and leg motor functions after complete paralysis. Nat Med. 2022 Feb;28(2):260-271. doi: 10.1038/s41591-021-01663-5. Epub 2022 Feb 7. PMID 35132264
- [Background] Lorach H, Galvez A, Spagnolo V, Martel F, Karakas S, Intering N, Vat M, Faivre O, Harte C, Komi S, Ravier J, Collin T, Coquoz L, Sakr I, Baaklini E, Hernandez-Charpak SD, Dumont G, Buschman R, Buse N, Denison T, van Nes I, Asboth L, Watrin A, Struber L, Sauter-Starace F, Langar L, Auboiroux V, Carda S, Chabardes S, Aksenova T, Demesmaeker R, Charvet G, Bloch J, Courtine G. Walking naturally after spinal cord injury using a brain-spine interface. Nature. 2023 Jun;618(7963):126-133. doi: 10.1038/s41586-023-06094-5. Epub 2023 May 24. PMID 37225984
- [Background] Liu P, Cheng Y, Xu Z, Li X, Chen Z, Duan W. Spatiotemporal spinal cord stimulation with real-time triggering exoskeleton restores walking capability: a case report. Ann Clin Transl Neurol. 2025 Mar;12(3):659-665. doi: 10.1002/acn3.52281. Epub 2024 Dec 15. PMID 39675019